CLINICAL TRIAL: NCT02874976
Title: Phototherapy Applied in Combination With Aerobic Training: Evaluation of Different Irradiation Protocols
Brief Title: Phototherapy Applied in Combination With Aerobic Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Larissa Aline Santos, Study Diretor, Ernesto Leal Junior, PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LSantos, UniNove
Record Dates: First submitted 2016-07-18; First posted 2016-08-22 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Excessive Physical Exercise, Unspecified
Keywords: sedentary lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Experimental: Group A (Experimental): Active and Active Phototherapy The phototherapy was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group A, received program 1 before aerobic training, and the same program 1 after training
  Interventions: Device: Active and Active Phototherapy; Device: Active and Placebo Phototherapy; Device: Placebo and active Phototherapy; Device: Placebo and Placebo Phototherapy
- Experimental: Group B (Experimental): Active and Placebo Phototherapy The phototherapy was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group B, received program 1 before aerobic training, and program 2 after training.
  Interventions: Device: Active and Active Phototherapy; Device: Active and Placebo Phototherapy; Device: Placebo and active Phototherapy; Device: Placebo and Placebo Phototherapy
- Experimental: Group C (Experimental): Placebo and Active Phototherapy The phototherapy was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group C, received program 2 before aerobic training, and program 1 after training.
  Interventions: Device: Active and Active Phototherapy; Device: Active and Placebo Phototherapy; Device: Placebo and active Phototherapy; Device: Placebo and Placebo Phototherapy
- Experimental: Group D (Experimental): Placebo and Placebo Phototherapy The phototherapy was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group B, received program 2 before strength training, and the same program 2 after training.
  Interventions: Device: Active and Active Phototherapy; Device: Active and Placebo Phototherapy; Device: Placebo and active Phototherapy; Device: Placebo and Placebo Phototherapy

INTERVENTIONS:
Device: Active and Active Phototherapy — Participants performed a aerobic training. Ninety-six subjects practice a regular aerobic exercise program on a treadmill was applied 3 times a week for 12 weeks,each session lasting 30 minutes, ranging between 70-80 % of maximum heart rate intensity and the evaluations are done monthly through a maximum progressive exercise protocol. Phototherapy, active or placebo, were applied in 9 different points of quadriceps,6 points in the posterior thigh and two points in the gastrocnemius muscle, depending the group randomized, before and after each training session.
Device: Active and Placebo Phototherapy — Participants performed a aerobic training. Ninety-six subjects practice a regular aerobic exercise program on a treadmill was applied 3 times a week for 12 weeks,each session lasting 30 minutes, ranging between 70-80 % of maximum heart rate intensity and the evaluations are done monthly through a maximum progressive exercise protocol. Phototherapy, active or placebo, were applied in 9 different points of quadriceps,6 points in the posterior thigh and two points in the gastrocnemius muscle, depending the group randomized, before and after each training session.
Device: Placebo and active Phototherapy — Participants performed a aerobic training. Ninety-six subjects practice a regular aerobic exercise program on a treadmill was applied 3 times a week for 12 weeks,each session lasting 30 minutes, ranging between 70-80 % of maximum heart rate intensity and the evaluations are done monthly through a maximum progressive exercise protocol. Phototherapy, active or placebo, were applied in 9 different points of quadriceps,6 points in the posterior thigh and two points in the gastrocnemius muscle, depending the group randomized, before and after each training session.
Device: Placebo and Placebo Phototherapy — Participants performed a aerobic training. Ninety-six subjects practice a regular aerobic exercise program on a treadmill was applied 3 times a week for 12 weeks,each session lasting 30 minutes, ranging between 70-80 % of maximum heart rate intensity and the evaluations are done monthly through a maximum progressive exercise protocol. Phototherapy, active or placebo, were applied in 9 different points of quadriceps,6 points in the posterior thigh and two points in the gastrocnemius muscle, depending the group randomized, before and after each training session.

SUMMARY:
Interventional

DETAILED DESCRIPTION:
Allocation: Randomized Endpoint Classification: Safety/Efficacy Study Intervention Model: Single Group Assignment Masking: Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor) Primary Purpose: Supportive Care

ELIGIBILITY:
Inclusion Criteria:

* There were included in the study
* healthy individuals,
* aged between 18 and 35 years old,
* presenting no history of musculoskeletal injury.
* that are not making use of pharmacological agents and / or nutritional supplements, and that have at least 80% of attendance to training.

Exclusion Criteria:

* present some musculoskeletal injury during the study
* cardiac ou pulmonary disease severe

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time until exhaustion | change from baseline in the time until exhaustion at 12 weeks
  ergoespirometry

SECONDARY OUTCOMES:
Maximum consumption of oxygen VO2 | change from baseline in the Maximum consumption of oxygen at 12 weeks
  ergoespirometry
Body fat | change from baseline in the body fat at 12 weeks
  skinfold

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Leal-Junior, PHD, Study Chair — Study Principal Investigator - Universidade Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No